CLINICAL TRIAL: NCT04533724
Title: Study on the Gut Microbial Mechanism of Negative Symptoms of Schizophrenia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020LQY
Record Dates: First submitted 2020-08-22; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Negative Symptom; Schizophrenia; Amisulpride; Gut Microbiomes
Keywords: Gut microbiota-brain axis; Negative symptom; Schizophrenia; Amisulpride
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Recruit 30 outpatient/inpatient schizophrenia patients (dominant negative symptoms) in Shanghai Mental Health Center .
  Interventions: Drug: Amisulpride
- Healthy control group (No Intervention): 15 cases of normal healthy people (control group) with similar eating habits and ages in the same region were matched with study group.

INTERVENTIONS:
Drug: Amisulpride — The amisulpride treatment group was given amisulpride tablets. The dose: the initial dose was 50 mg/d. The doctor titrated the dose to the therapeutic amount within 1 to 2 weeks according to the patient's condition. The maximum dose was 300 mg/d, taken with a single meal. Observe for 8 weeks.
  Arms: Study group

SUMMARY:
Negative symptoms are one of the five-dimensional symptoms of patients with schizophrenia, and medications are not effective in treating negative symptoms. The mechanism of negative symptoms of schizophrenia is unknown, which may be related to insufficient dopamine function of the prefrontal cortex. Amisulpride is a D2/D3 receptor antagonist, which can improve negative symptoms. Intestinal microbes are related to central nervous system mental diseases. Animal studies have found that changes in the intestinal microflora are related to schizophrenia. Clinical studies have found that the gut microbes of patients with schizophrenia are different from those of normal healthy people. Therefore, we are trying to discover the changes of gut microbes in patients with effective amisulpride treatment, and to improve the negative symptoms of schizophrenia patients through the intestinal immune system. The mechanism of brain relationship provides direction, and also provides a new way for the drug treatment of negative symptoms.

DETAILED DESCRIPTION:
Negative symptoms are one of the five-dimensional symptoms of patients with schizophrenia. Drug treatment of negative symptoms is not effective. Even if the positive symptoms are relieved, the negative symptoms continue to exist, which seriously affects the personal family social function and is an important risk factor for poor prognosis. The mechanism of negative symptoms of schizophrenia is unknown, which may be related to insufficient dopamine function of the prefrontal cortex, but the pathogenesis is still not fully explained. Amisulpride is a D2/D3 receptor antagonist, which can improve negative symptoms, but the mechanism is not clear. Intestinal microbes are related to central nervous system psychiatric diseases, and intestinal flora imbalance may be an important cause of autism, anxiety, depression, schizophrenia and other mental and psychological diseases. Under pathological conditions, when the intestinal microbiome is disturbed or the intestinal mucosal barrier is destroyed, microbial-related molecules stimulate macrophages and dendritic cells to produce pro-inflammatory cytokines, which in turn activate adaptive immune cells, leading to the destruction of immune homeostasis and enteric nerves The system can also interact with the central nervous system through the brain-gut axis. Intestinal microbes may also influence the occurrence of mental illness through metabolites. Animal studies have found that changes in the intestinal microflora are related to schizophrenia. Clinical studies have found that the gut microbes of patients with schizophrenia are different from those of normal healthy people. Therefore, we are trying to discover the changes of gut microbes in patients with effective amisulpride treatment, and to improve the negative symptoms of schizophrenia patients through the intestinal immune system. The mechanism of brain relationship provides direction, and also provides a new way for the drug treatment of negative symptoms. This study intends to select 30 patients with schizophrenia with dominant negative symptoms (study group) and 15 healthy people with similar living environment (control group), and the study group will be treated with amisulpride (flexible treatment), negative symptom factor The score reduction rate reached 20% for the effective group. Followed up for 8 weeks, fresh stool samples were collected at the baseline, 2, 4, and 8 weekends for 16S rRNA sequencing and short-chain fatty acid detection, and whole blood samples for immune factors (IL-1β, IL-6, IL-10, TNF) -α) Test to assess the negative symptom factor scores of PANSS, CDSS, CGI, TESS, SAS, and Barnes akathisia, and evaluate the patient's negative symptoms, depressive symptoms, efficacy and adverse reactions in turn. Comparing the differences in the intestinal microflora of the two groups at baseline, the correlation between the changes of the intestinal microflora of the effective group of amisulpride and the immune factors and negative symptoms. To understand the pathogenesis of schizophrenia patients with dominant negative symptoms through the gut microbiota-brain axis.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old, Han nationality, no gender limit;
* Meet the diagnostic criteria of "Schizophrenia" in the American Diagnostic Standards for Mental Disorders (DSM-V);
* The first attack, no antipsychotic drugs have been used in the past six months;
* The PANSS negative symptom subscale has at least 3 items with 4 points and above or at least two items with 5 points and above, and the positive symptoms score is less than 19 points;
* The negative symptom score is at least 6 points or more higher than the positive symptom score;
* The cultural, social and educational background is sufficient to understand informed consent and research content.

Exclusion Criteria:

* 1.Combined with DSM-V diagnosis other than schizophrenia;
* .G6≥4 points in PANSS, or CDSS≥6 points;
* .SAS Side Reaction Scale> 3 points;
* Organic diseases of the central nervous system;
* In the past two months, there were people who were dependent or abused on alcohol or other substances, which caused significant impairment of social and cognitive function;
* In the past year, there have been major life events such as widowhood;
* Serious suicide attempts;
* .The current patient's severe and unstable physical disease;
* .Pregnant and lactating women;
* Have a history of antibiotic use of more than 3 days within 3 months;
* Use probiotics (lactic acid products, etc.) for more than 3 days within 3 months;
* Type 1 diabetes and severe diabetes complications;
* .Digestive system diseases such as gastrointestinal inflammation, acute or chronic hepatitis;
* .Severe organ diseases, such as cancer, coronary heart disease, myocardial infarction, cerebral hemorrhage;
* .Have infectious diseases, such as tuberculosis, AIDS;
* Drug treatment of cholecystitis, peptic ulcer, urinary tract infection, acute nephritis, cystitis or hyperthyroidism.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The change of intestinal microbial flora | 12 weeks
  The main evaluation index is the difference between the change of intestinal microbial flora in the study group and the control group before and after treatment.

SECONDARY OUTCOMES:
PANSS negative symptom scale score reduction rate | 12 weeks
  The secondary evaluation index is the PANSS negative symptom scale score reduction rate ≥ 20%

CONTACTS AND LOCATIONS:
Overall Officials: Qinyu Lv, Principal Investigator — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine; Qi Zhang, Study Chair — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine; Zhenghui Yi, Study Chair — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine; Congze Wang, Study Chair — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine; Huanling Zhang, Study Chair — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine; Xinxin Huang, Study Chair — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT04533724/Prot_SAP_000.pdf